CLINICAL TRIAL: NCT05316116
Title: A Pilot Study of Siltuximab in Large Granular Lymphocytic Leukemia (LGLL)
Brief Title: Siltuximab in Large Granular Lymphocytic Leukemia (LGLL)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of efficacy/futility
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: EUSA Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21035
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Large Granular Lymphocyte Leukemia
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic | interventions — siltuximab; Interleukin-6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Siltuximab (Experimental): Siltuximab will be given every 3 weeks, for between 18 and 36 weeks
  Interventions: Drug: Siltuximab

INTERVENTIONS:
Drug: Siltuximab — Siltuximab will be given on day 1 of each cycle. The dose will be 11 mg/kg given over 1 hour by intravenous infusion. Each cycle is three weeks (+-3 days).
  Other Names: Interleukin-6

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of siltuximab for participants being treated for large granular lymphocytic leukemia (LGLL).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged >/= 18.
* Meet the diagnosis criteria of LGLL as below:
* a. For a patient with treatment-naive LGLL, peripheral blood needs to have CD3+ CD57+ cells >400/mm³ or CD8+ cells >650/mm³, and, evidence for clonal T cell receptor gamma or beta gene rearrangement by PCR needs to be detected in either peripheral blood or bone marrow.
* b. For patients with an established diagnosis of LGLL who have been previously treated, multicolor flow cytometry should identify a residual CD3+CD57+CD8+ LGLL population in peripheral blood or bone marrow, and, evidence for clonal T cell receptor gamma or beta gene rearrangement by PCR needs to be detected in either peripheral blood or bone marrow. There is no requirement that peripheral blood absolute clonal CD3+ CD57+ or CD8+ LGLL populations need to reach predetermined minimal value for eligibility since immunosuppressive therapy can significantly decrease LGLL cell count without any impact on neutropenia, anemia or thrombocytopenia which are major causes of morbidity and mortality
* Has at least one of the indications for treatment:

  1. severe neutropenia less than 500/mm³, OR
  2. neutropenia associated with recurrent infection, OR
  3. symptomatic anemia with Hemoglobin < 9 g/dL, OR
  4. transfusion-dependent anemia with transfusion needs >= 1 u per month, OR
  5. severe thrombocytopenia <20,000/mm³, OR
  6. thrombocytopenia <50,000/mm³ with bleeding.
* Participant can be treatment-naïve or previously treated for LGLL.
* Participant currently receiving therapy must have a wash-out period of ≥ 30 days or 5 elimination half-lives, whichever is longer, prior to study drug administration.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Creatinine clearance (CLCr) ≥15 mL/min.
* If a participant has chronic liver disease, Child-Pugh score needs to be either A or B.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to study drug infusion and agreement to use highly effective contraception during study participation and for an additional 3 months after the last dose of study drug.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during study participation and for an additional 3 months after the last dose of study drug. Men must agree to not donate sperm during the same period.

Exclusion Criteria:

* Any active infection requiring systemic therapy, including viral infections such as HIV, Hepatitis B, and/or Hepatitis C.
* Current use of methotrexate, cyclophosphamide, or cyclosporine for any medical conditions.
* Has coexisting myelodysplastic syndrome (MDS).
* Elevated LGL due to viral infection.
* Pregnancy or lactation.
* Known severe allergic reactions to siltuximab.
* At increased risk for Gastrointestinal (GI) perforation, in the opinion of the study investigator.
* Received live vaccine 30 days prior to study drug administration or Intend to receive live vaccine during treatment period and within 3 months after last dose of study drug.
* Rheumatological conditions such as rheumatoid arthritis (RA) are not exclusion criteria for the study.
* Coexisting hematological conditions such as autoimmune hematological anemia (AIHA) or immune thrombocytopenia (ITP) are not automatic exclusion criteria but will be at discretion of study investigator.
* Previous or concurrent malignancies not considered cured, except inactive non-melanoma skin cancer, in situ carcinoma of the cervix, early-stage prostate cancer, or other cancer deemed clinically insignificant by the Investigator.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the study Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 30 months
  Overall response rate is defined as the rate of achieving best response of CR or PR, and will be summarized for participants who have received any dose of study drug

SECONDARY OUTCOMES:
Complete Response Rate (CR) | Up to 30 months
  CR rate is defined as the percentage of patients achieving best response of CR.
Time to Response (TTR) | Up to 30 months
  TTR is defined as time from first dose of study drug to time of meeting criteria for CR or PR, whichever comes first.
Duration of Response (DOR) | Up to 30 months
  Duration of Response is defined as time from achieving either CR or PR, whichever comes first, to time of progression or starting another LGLL treatment, whichever comes first.
Duration of Complete Response | Up to 30 months
  Duration of CR is defined as time from achieving CR to time of progression or starting another LGLL treatment, whichever comes first.
Time to Complete Response | Up to 30 months
  Time to CR is defined as time from first dose of study drug to time of CR
Duration of Complete Response with Normalization of PB LGL Count | Up to 30 months
  Rate of CR with normalization of PB LGL count is defined as meeting criteria for CR AND a normal PB LGL count ( <400/mm³ CD3+CD57+ cells or <650/mm³ CD8+ T cells in PB).
Progression Free Survival | Up to 30 months
  PFS is defined as time from first dose of study drug to time of disease progression or starting another LGLL treatment, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Lubomir Sokol, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinicaltrialssearch?DiseaseSite=&q=21035